CLINICAL TRIAL: NCT03463226
Title: Hormonal Anabolic Deficiency Associated With Neurovascular Alterations Predict Poor Prognosis in Male Patients With Heart Failure
Brief Title: Effects of Hormonal Anabolic Deficiency and Neurovascular Alterations on Mortality in Male Patients With Heart Failure
Acronym: TestoHF
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maria Janieire de Nazaré Nunes Alves, PhD, University of Sao Paulo General Hospital
Other Study IDs: AnabolicHormonesPrognosis
Record Dates: First submitted 2018-03-01; First posted 2018-03-13 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: Testosterone Deficiency; Sympathetic overactivity; Exercise Intolerance
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low testosterone: Patients with HF and testosterone deficiency.
  * Cardiopulmonary exercise test
  * Muscle Sympathetic Nerve Activity
  * Dual-energy X-ray absorptiometry
  * Venous occlusion plethysmography
  * Blood sample collection
  * Dynamometers for Handgrip Strength
  Interventions: Diagnostic Test: Cardiopulmonary exercise test; Diagnostic Test: Muscle Sympathetic Nerve Activity; Diagnostic Test: Dual-energy X-ray absorptiometry; Diagnostic Test: Venous occlusion plethysmography; Diagnostic Test: Blood sample collection; Diagnostic Test: Dynamometers for Handgrip Strength
- Normal testosterone: Patients with HF and normal plasma levels of testosterone.
  * Cardiopulmonary exercise test
  * Muscle Sympathetic Nerve Activity
  * Dual-energy X-ray absorptiometry
  * Venous occlusion plethysmography
  * Blood sample collection
  * Dynamometers for Handgrip Strength
  Interventions: Diagnostic Test: Cardiopulmonary exercise test; Diagnostic Test: Muscle Sympathetic Nerve Activity; Diagnostic Test: Dual-energy X-ray absorptiometry; Diagnostic Test: Venous occlusion plethysmography; Diagnostic Test: Blood sample collection; Diagnostic Test: Dynamometers for Handgrip Strength

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — Oxygen consumption (VO2) and carbon dioxide output (VCO2) were measured by means of gas exchange on a breath-by-breath basis. The patients were initially monitored for 2 minutes at rest when seated on the ergometer, after that they were instructed to pedal at a pace of 60-70 rpm and the completion of the test occurred when, in spite of verbal encouragement, the patient reached maximal volitional fatigue.
Diagnostic Test: Muscle Sympathetic Nerve Activity — Multiunit post-ganglionic muscle sympathetic nerve recordings were made using a tungsten microelectrode placed in the peroneal nerve near the fibular head. Nerve signals were amplified by a factor of 50,000 to 100,000 and band-pass filtered (700 to 2000 Hz). For recording and analysis, nerve activity was rectified and integrated (time constant 0.1 seconds) to obtain a mean voltage display of sympathetic nerve activity.
Diagnostic Test: Dual-energy X-ray absorptiometry — Dual-energy X-ray absorptiometry (DXA) scan was used to measure total lean mass, body fat and bone mineral content.
Diagnostic Test: Venous occlusion plethysmography — Venous occlusion plethysmography was used to assess non-invasively blood flow.
Diagnostic Test: Blood sample collection — Blood samples were drawn in the morning after 12h overnight fasting.
Diagnostic Test: Dynamometers for Handgrip Strength — Muscle strength was assessed by handgrip dynamometer using the mean value of three attempts.

SUMMARY:
Heart failure (HF) has been associated with chronic deleterious effects on skeletal muscle, endocrine system, vasculature and sympathetic nervous system. These alterations have a significant impact on quality of life, leading to a reduction in functional capacity and limited symptoms, which involve dyspnea and fatigue. The investigators tested the hypothesis that hormonal anabolic deficiency associated with neurovascular alterations may worsen the prognosis of patients with heart failure.

DETAILED DESCRIPTION:
One hundred and fifty six patients have been enrolled so far. Methods were as described below:

* Muscle sympathetic nerve activity (MSNA) was directly recorded from the peroneal nerve using the microneurography technique ;
* All patients underwent symptom-limited cardiopulmonary exercise test performed on a cycle ergometer, using a ramp protocol with workload increments of 5 or 10 Watts per minute;
* Body composition measurements were performed using dual-energy X-ray absorptiometry (DXA);
* Muscle strength was assessed by handgrip dynamometer using the mean value of three attempts;
* Blood samples were drawn in the morning after 12h overnight fasting. The laboratory tests included B-type natriuretic peptide (BNP; pg/mL) plasma level, serum sodium (mEq/L), serum potassium (mEq/L), creatinine (mg/dL), haemoglobin level (g/dL), high-sensitivity C-reactive protein (CRP; mg/L), lipid profile (triglyceride, total cholesterol, high-density lipoprotein, and low-density lipoprotein; mg/dL), and fasting glucose (mg/dL). Blood sample to assess hormone plasma levels were also drawn at the same time: total testosterone (TT), free testosterone (FT), sex hormone binding globulin (SHBG), dehydroepiandrosterone sulfate (DHEAS), luteinizing hormone (LH), follicle-stimulating hormone (FSH), thyroid stimulating hormone (TSH) and insulin-like growth factor 1 (IGF1).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years old;
* at least1 year of diagnosed HF;
* left ventricular ejection fraction (LVEF) lower than 40% measured by echocardiography;
* non-ischaemic and ischaemic aetiologies;
* compensated HF with optimal medication for at least 3 months prior the study;
* New York Heart Association (NYHA) class of I to IV.

Exclusion Criteria:

* patients with autonomic diabetic neuropathy;
* patients with chronic renal failure with haemodialysis;
* heart transplantation;
* presence of pacemaker;
* patients with muscular dystrophy (i.e. Duchenne muscular dystrophy);
* patients submitted to any hormonal treatment;
* history of cancer;
* ongoing infection;
* myocardial infarction with percutaneous coronary intervention or revascularization 6 months prior to the study entry.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure recruited at Clinical Unit of Myocardiopathy at General Hospital of the University of São Paulo Medical School (UNCAR/HC-FMUSP).
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Impact of testosterone deficiency on mortality | 2 years
  Blood sample was collected in the morning (between 8:00-10:00 a.m.) after 12 hours fasting.
Impact of muscle sympathetic nerve activity on mortality | 2 years
  Microneurography was used to assess the sympathetic nervous system.
Impact of neurovascular alterations on mortality | 2 years
  Venous occlusion pletysmography was used to evaluate vasodilation.

SECONDARY OUTCOMES:
Impact of testosterone deficiency on body composition | 2 years
  Body composition measurements were performed using dual-energy X-ray absorptiometry.
Impact of testosterone deficiency on functional capacity | 2 years
  All patients underwent symptom-limited cardiopulmonary exercise test to measure functional capacity.
Impact of testosterone deficiency on strength | 2 years
  Muscle strength was assessed by handgrip dynamometer using the mean value of three attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Janieire de Nazaré Nunes Alves, PhD, Principal Investigator — InCor Heart Institute
Locations (1):
- Instituto do Coração do Hospital da Clínicas da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No